CLINICAL TRIAL: NCT05049694
Title: Clinical and Radiographic Performance of Preformed Zirconia Crowns and Stainless-Steel Crowns in Permanent First Molars: 18-Month Results of a Prospective, Randomized Trial
Brief Title: Success of Zirconia and Stainless Steel Crowns for Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zafer Cavit Cehreli, DDS, PhD, Prof.Dr., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: posterior permanent crown rest
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Caries Active; Dentin, Carious
Keywords: zirconia crowns; stainless steel crowns; dental caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zirconia crowns (Experimental): esthetic crowns for capping permanent molars with caries
  Interventions: Device: zirconia crowns
- stainless steel crowns (Experimental): stainless steel crowns for capping permanent molars with caries
  Interventions: Device: stainless steel crowns

INTERVENTIONS:
Device: zirconia crowns — esthetic crowns for capping permanent molars with caries
  Arms: zirconia crowns
Device: stainless steel crowns — stainless steel crowns for capping permanent molars with caries
  Arms: stainless steel crowns

SUMMARY:
The purpose of this study is to evaluate and compare the clinical and radiographic performance of zirconia and stainless steel crowns on permanent molar

DETAILED DESCRIPTION:
Zirconia and stainless steel crowns will be placed on at least two permanent molars, in a split mouth design. 100 patients will be included in the study. The teeth will be randomized into two groups according to the crown type.

Group 1: Zirconia crown 2: Stainless steel crown. Plaque index, gingival index, crown retention, presence of restoration failure, gingival margin extension and pulpal health of the teeth will be clinically evaluated at baseline and 1., 6., 12., 18., 24. months. The restorations will be evaluated radiographically at 6., 12. and 18. months. Intra-oral photos will be taken directly after treatment and at control appointments.

The data will be analysed statistically using Fisher's Exact Test and pearson's chi-square test; and Log-rank and the Kaplan-Meier will be used to estimate survival percentages.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parent of the patients who accept to participate and sign the informed consent
* Patients who have at least two permanent molars with caries that require crown restoration
* Patients that have good cooperation to the procedure

Exclusion Criteria:

* Patients and parent of the patients who don't accept to participate and sign the informed consent
* Teeth that doesn't have opposing permanent molars
* Patients who have bruxism or deep-bite
* Patient who are allergic to nickel

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of zirconia and stainless steel crowns that showed successful retention over two years | 2 years
  Long-term clinical success of zirconia and stainless steel crowns placed on permanent molars

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Geduk N, Ozdemir M, Erbas Unverdi G, Ballikaya E, Cehreli ZC. Clinical and radiographic performance of preformed zirconia crowns and stainless-steel crowns in permanent first molars: 18-month results of a prospective, randomized trial. BMC Oral Health. 2023 Nov 3;23(1):828. doi: 10.1186/s12903-023-03501-1. PMID 37924021